CLINICAL TRIAL: NCT02291289
Title: A Multi-Centre Randomised Clinical Trial of Biomarker-Driven Maintenance Treatment for First-Line Metastatic Colorectal Cancer (MODUL)
Brief Title: A Study of Biomarker-Driven Therapy in Metastatic Colorectal Cancer (mCRC)
Acronym: MODUL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO29112; 2014-001017-61 (EudraCT Number)
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Capecitabine; atezolizumab; Vemurafenib; Bevacizumab; Trastuzumab; pertuzumab; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- Cohort 1: Induction Phase (IP) (Other): Includes participants with v-raf murine sarcoma viral oncogene homolog B1 mutation positive (BRAFmut)/human epidermal growth factor receptor 2 negative (HER2-)/microsatellite stable (MSS)/rat sarcoma wild type (RASwt). All participants will receive either eight 2-week cycles of 5-fluorouracil (5-FU)/ leucovorin calcium (LV) and oxaliplatin (FOLFOX) in combination with bevacizumab, or six 2-week cycles of FOLFOX in combination with bevacizumab, followed by two 2-week cycles of 5-FU/LV with bevacizumab.
  Interventions: Drug: FOLFOX induction regimen; Drug: Bevacizumab; Drug: 5-FU/LV
- Cohort 2 (IP) (Other): Includes participants with BRAFwt. All participants will receive either eight 2-week cycles of 5-fluorouracil (5-FU)/ leucovorin calcium (LV) and oxaliplatin (FOLFOX) in combination with bevacizumab, or six 2-week cycles of FOLFOX in combination with bevacizumab, followed by two 2-week cycles of 5-FU/LV with bevacizumab.
  Interventions: Drug: FOLFOX induction regimen; Drug: Bevacizumab; Drug: 5-FU/LV
- Cohort 3 (IP) (Other): Includes participants with human epidermal growth factor receptor 2 positive (HER2+). All participants will receive either eight 2-week cycles of 5-fluorouracil (5-FU)/ leucovorin calcium (LV) and oxaliplatin (FOLFOX) in combination with bevacizumab, or six 2-week cycles of FOLFOX in combination with bevacizumab, followed by two 2-week cycles of 5-FU/LV with bevacizumab.
  Interventions: Drug: FOLFOX induction regimen; Drug: Bevacizumab; Drug: 5-FU/LV
- Cohort 4 (IP) (Other): Includes participants with HER2-/high microsatellite instability (MSI-H); HER2-/MSS/v-raf murine sarcoma viral oncogene homolog B1 wild type (BRAFwt); HER2-/MSS/BRAFmut/rat sarcoma mutation positive (RASmut). All participants will receive either eight 2-week cycles of 5-fluorouracil (5-FU)/ leucovorin calcium (LV) and oxaliplatin (FOLFOX) in combination with bevacizumab, or six 2-week cycles of FOLFOX in combination with bevacizumab, followed by two 2-week cycles of 5-FU/LV with bevacizumab.
  Interventions: Drug: FOLFOX induction regimen; Drug: Bevacizumab; Drug: 5-FU/LV
- Cohort 1 (Maintenance Phase[MP]):5-FU/LV,cetuximab,vemurafenib (Experimental): Participants with v-raf murine sarcoma viral oncogene homolog B1 mutation positive (BRAFmut)/human epidermal growth factor receptor 2 negative (HER2-)/microsatellite stable (MSS)/rat sarcoma wild type (RASwt) will receive 1600-2400 milligrams per square meter (mg/m^2) 5-FU via 46-hour intravenous (IV) infusion in combination with 400 mg/m^2 LV via 2-hour infusion on Day 1 of every 2-week cycle with 500 mg/m^2 cetuximab via infusion on Day 1 of every 2-week cycle and 960 milligrams (mg) vemurafenib twice daily (BID) by mouth.
  Interventions: Drug: Cetuximab; Drug: Vemurafenib; Drug: 5-FU/LV
- Cohort 1 Control (MP): 5-FU/LV or capecitabin, bevacizumab (Active Comparator): Per Investigator discretion, participants will receive fluoropyrimidine (5-FU/LV or capecitabine) at a dose and schedule per the Investigator's discretion in accordance with locally approved prescribing information and 5 mg/kg bevacizumab via 1-30 minute IV on Day 1 of every 2-week cycle.
  Interventions: Drug: Fluoropyrimidine (5-FU/LV or capecitabine); Drug: Bevacizumab
- Cohort 2 (MP):5-FU/LV or capecitabine,bevacizumab,atezolizumab (Experimental): Participants with BRAFwt will receive fluoropyrimidine (1600-2400 mg/m^2 5-FU via 46-hour IV infusion in combination with 400 mg/m^2 LV via 2-hour infusion on Day 1 of every 2-week cycle or 1000 mg/m^2 twice-daily capecitabine BID by mouth on Days 1-14 every 2 weeks followed by a 1-week break) with 5 milligrams per kilogram (mg/kg) bevacizumab via 15-30 minute IV infusion on Day 1 of every 2-week cycle and 800 mg atezolizumab via 60-minute IV infusion on Day 1 of every 2-week cycle.
  Interventions: Drug: Fluoropyrimidine (5-FU/LV or capecitabine); Drug: Atezolizumab; Drug: Bevacizumab
- Cohort 2 Control (MP): 5-FU/LV or capecitabin, bevacizumab (Active Comparator): Per Investigator discretion, participants will receive fluoropyrimidine (5-FU/LV or capecitabine) at a dose and schedule per the Investigator's discretion in accordance with locally approved prescribing information and 5 mg/kg bevacizumab via 1-30 minute IV on Day 1 of every 2-week cycle.
  Interventions: Drug: Fluoropyrimidine (5-FU/LV or capecitabine); Drug: Bevacizumab
- Cohort 3 (MP): capecitabine,trastuzumab,pertuzumab (Experimental): Participants with human epidermal growth factor receptor 2 positive (HER2+) will receive 1000 mg/m^2 twice-daily capecitabine BID by mouth on Days 1-14 every 2 weeks followed by a 1-week break with trastuzumab by IV infusion on Day 1 of every 3-week treatment cycle at an initial loading dose of 8 mg/kg followed by 6 mg/kg for subsequent doses, and pertuzumab by IV infusion on Day 1 of each 3-week treatment cycle at an initial fixed loading dose of 840 mg followed by 420 mg for subsequent doses.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Capecitabine
- Cohort 3 Control (MP): 5-FU/LV or capecitabin, bevacizumab (Active Comparator): Per Investigator discretion, participants will receive fluoropyrimidine (5-FU/LV or capecitabine) at a dose and schedule per the Investigator's discretion in accordance with locally approved prescribing information and 5 mg/kg bevacizumab via 1-30 minute IV on Day 1 of every 2-week cycle.
  Interventions: Drug: Fluoropyrimidine (5-FU/LV or capecitabine); Drug: Bevacizumab
- Cohort 4 (MP): Cobimetinib,atezolizumab (Experimental): Participants with HER2-/high microsatellite instability (MSI-H); HER2-/MSS/v-raf murine sarcoma viral oncogene homolog B1 wild type (BRAFwt); HER2-/MSS/BRAFmut/rat sarcoma mutation positive (RASmut) will receive 60 mg cobimetinib orally for 3 weeks followed by a 1-week treatment break and atezolizumab at a fixed dose of 840 mg via 60-minute IV infusion on Day 1 of every 2-week cycle.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib
- Cohort 4 Control (MP): 5-FU/LV or capecitabin, bevacizumab (Active Comparator): Per Investigator discretion, participants will receive fluoropyrimidine (5-FU/LV or capecitabine) at a dose and schedule per the Investigator's discretion in accordance with locally approved prescribing information and 5 mg/kg bevacizumab via 1-30 minute IV on Day 1 of every 2-week cycle.
  Interventions: Drug: Fluoropyrimidine (5-FU/LV or capecitabine); Drug: Bevacizumab
- Early Progressing BRAFmut Cohort (Other): BRAFmut participants experiencing early disease progression during induction treatment will have the option of proceeding immediately to receive second-line treatment with 5-FU/LV, cetuximab and vemurafenib if their primary tumor is MSS, or with a fluoropyrimidine (5-FU/LV or capecitabine), bevacizumab, and atezolizumab if their primary tumor is MSI-H. This cohort will be followed for adverse events during the study, but is not part of the Maintenance Phase study objectives.
  Interventions: Drug: Cetuximab; Drug: Fluoropyrimidine (5-FU/LV or capecitabine); Drug: Atezolizumab; Drug: Vemurafenib; Drug: Bevacizumab; Drug: 5-FU/LV

INTERVENTIONS:
Drug: Cetuximab — 500 mg/m^2 via IV infusion on Day 1 of every 2-week cycle
  Arms: Cohort 1 (Maintenance Phase[MP]):5-FU/LV,cetuximab,vemurafenib; Early Progressing BRAFmut Cohort
Drug: FOLFOX induction regimen — Administered per the Investigator's discretion in accordance with locally approved prescribing information.
  Arms: Cohort 1: Induction Phase (IP); Cohort 2 (IP); Cohort 3 (IP); Cohort 4 (IP)
Drug: Fluoropyrimidine (5-FU/LV or capecitabine) — Per Investigator's discretion: 5-FU 1600-2400 mg/m^2 administered via 46-hour IV infusion on Day 1 of every 2-week cycle and LV 400 mg/m^2 administered via a 2-hour infusion on Day 1 every 2 weeks or 1000 mg/m^2 twice-daily capecitabine (BID) by mouth given days 1-14 every 2 weeks. The chosen fluoropyrimidine should be administered in accordance with local prescribing information.
  Arms: Cohort 1 Control (MP): 5-FU/LV or capecitabin, bevacizumab; Cohort 2 (MP):5-FU/LV or capecitabine,bevacizumab,atezolizumab; Cohort 2 Control (MP): 5-FU/LV or capecitabin, bevacizumab; Cohort 3 Control (MP): 5-FU/LV or capecitabin, bevacizumab; Cohort 4 Control (MP): 5-FU/LV or capecitabin, bevacizumab; Early Progressing BRAFmut Cohort
Drug: Atezolizumab — 800 mg atezolizumab via 60-minute IV infusion on Day 1 of every 2-week cycle, or a fixed dose of 840 mg
  Other Names: MPDL3280A, RO5541267
  Arms: Cohort 2 (MP):5-FU/LV or capecitabine,bevacizumab,atezolizumab; Cohort 4 (MP): Cobimetinib,atezolizumab; Early Progressing BRAFmut Cohort
Drug: Vemurafenib — 960 mg vermurafenib BID by mouth
  Other Names: RO5185426
  Arms: Cohort 1 (Maintenance Phase[MP]):5-FU/LV,cetuximab,vemurafenib; Early Progressing BRAFmut Cohort
Drug: Bevacizumab — 5 mg/kg bevacizumab via 15-30 minute IV infusion on Day 1 of every 2-week cycle per local prescribing information
  Other Names: RO4876646
  Arms: Cohort 1 Control (MP): 5-FU/LV or capecitabin, bevacizumab; Cohort 1: Induction Phase (IP); Cohort 2 (IP); Cohort 2 (MP):5-FU/LV or capecitabine,bevacizumab,atezolizumab; Cohort 2 Control (MP): 5-FU/LV or capecitabin, bevacizumab; Cohort 3 (IP); Cohort 3 Control (MP): 5-FU/LV or capecitabin, bevacizumab; Cohort 4 (IP); Cohort 4 Control (MP): 5-FU/LV or capecitabin, bevacizumab; Early Progressing BRAFmut Cohort
Drug: Trastuzumab — Initial loading dose of 8 mg/kg followed by 6 mg/kg for subsequent doses by IV infusion on Day 1 of every 3-week treatment cycle
  Other Names: RO0452317
  Arms: Cohort 3 (MP): capecitabine,trastuzumab,pertuzumab
Drug: Pertuzumab — Initial fixed loading dose of 840 mg followed by 420 mg for subsequent doses by IV infusion on Day 1 of each 3-week treatment cycle
  Other Names: RO4368451
  Arms: Cohort 3 (MP): capecitabine,trastuzumab,pertuzumab
Drug: Cobimetinib — 60 mg orally once daily for 3 weeks followed by a 1-week treatment break
  Other Names: RO5514041
  Arms: Cohort 4 (MP): Cobimetinib,atezolizumab
Drug: 5-FU/LV — 1600-2400 mg/m^2 5-FU via 46-hour IV infusion in combination with 400 mg/m^2 LV via 2-hour infusion on Day 1 of every 2-week cycle until disease progression per the Investigator's assessment using modified Response Evaluation Criteria in Solid Tumors or death from any cause, whichever occurs first. The fluoropyrimidine should be administered in accordance with local prescribing information.
  Arms: Cohort 1 (Maintenance Phase[MP]):5-FU/LV,cetuximab,vemurafenib; Cohort 1: Induction Phase (IP); Cohort 2 (IP); Cohort 3 (IP); Cohort 4 (IP); Early Progressing BRAFmut Cohort
Drug: Capecitabine — 1000 mg/m^2 twice-daily capecitabine (BID) by mouth given days 1-14 every 2 weeks. The fluoropyrimidine should be administered in accordance with local prescribing information.
  Arms: Cohort 3 (MP): capecitabine,trastuzumab,pertuzumab

SUMMARY:
This randomized, multi-center, active-controlled, open-label, parallel-group study will investigate the efficacy and safety of biomarker-driven maintenance treatment for first-line mCRC. Participants with mCRC are eligible for entry and cannot have received any prior chemotherapy in the metastatic setting. The entire study duration is anticipated to be approximately 7.5 years.

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS of less than or equal to (<=) 2
* At least 16 weeks of life expectancy at time of entry into the study
* Histologically confirmed colorectal cancer (CRC) with mCRC confirmed radiologically
* Measureable, unresectable disease according to RECIST 1.1
* No prior chemotherapy for CRC in the metastatic setting
* Archival tumor formalin-fixed paraffin-embedded tissue block from the primary tumor obtained at the time of the initial diagnosis is available
* Adequate hematological, liver and renal function
* Agreement to use highly effective measures of contraception

Exclusion Criteria for All Participants:

* Less than 6 months from completion of any prior neoadjuvant or adjuvant chemotherapy, radiotherapy
* Prior or current treatment with bevacizumab or any other anti-angiogenic drug (vascular endothelial growth factor or vascular endothelial growth factor receptor therapies or tyrosine kinase inhibitors)
* Current or recent (within 10 days of study enrollment) use of aspirin (more than [>] 325 milligrams per day [mg/day]), clopidogrel (> 75 mg/day), or current or recent (within 10 days prior to the start of study induction treatment) use of therapeutic oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes (prophylactic uses allowed)
* Active infection requiring intravenous antibiotics at the start of study induction treatment
* Previous or concurrent malignancy, except for adequately treated basal or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the participant has been disease-free for 5 years prior to study entry
* Inadequately controlled hypertension; prior history of hypertensive crisis or hypertensive encephalopathy
* Clinically significant (active) cardiovascular disease, for example cerebrovascular accidents <= 6 months prior to start of study induction treatment, myocardial infarction <= 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Functional Classification Grade II or greater congestive heart failure, or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of start of study induction treatment
* Active symptomatic or untreated central nervous system (CNS) metastases; CNS disease other than supratentorial or cerebellar metastases (in other words, patients with metastases to midbrain, pons, medulla or spinal cord are excluded); history of or known carcinomatous meningitis
* Known hypersensitivity to any component of any of the study induction or maintenance treatment medications
* Pregnancy or lactation

Exclusion Criteria for Participants in Cohort 1 (MP):

* Inability to swallow pills
* Refractory nausea and vomiting, malabsorption, external biliary shunt or significant bowel resection that would preclude adequate absorption
* History or presence of clinically significant ventricular or atrial dysrhythmias
* Corrected QT (QTc) interval >= 450 millisecond assessed within 3 weeks prior to randomization, long QT syndrome or, uncorrectable electrolyte abnormalities (including magnesium) or requirement for medicinal products known to prolong the QT interval
* ECOG PS > 2

Exclusion Criteria for Participants in Cohort 2 (MP):

* History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis at most recent chest imaging (computed tomography [CT] scan or magnetic resonance imaging [MRI])
* Positive test for human immunodeficiency virus (HIV)
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) at Screening
* Active tuberculosis
* Severe infection within 4 weeks prior to start of maintenance treatment including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia; has signs or symptoms of significant infection or has received oral or IV antibiotics within 2 weeks prior to start of maintenance treatment
* Administration of a live, attenuated vaccine within 4 weeks prior to start of maintenance treatment or anticipation that such a live attenuated vaccine will be required during the remainder of the study
* Prior treatment with cluster of differentiation (CD) 137 agonists, anti-cytotoxic T-lymphocyte-associated antigen (CTLA) 4, anti-programmed death-1 (PD-1), or anti-programmed death-ligand 1 (PD-L1) therapeutic antibody or pathway-targeting agents
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or five half-lives of the drug, whichever is longer, prior to start of maintenance treatment
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior to start of maintenance treatment, or anticipated requirement for systemic immunosuppressive medications during the remainder of the study
* If receiving receptor activator of nuclear factor kappa-B ligand (RANKL) inhibitor (for example, denosumab) and unwilling to adopt alternative treatment such as bisphosphonates while receiving atezolizumab

Exclusion Criteria for Participants in Cohort 3 (MP):

* Inability to swallow pills
* Left ventricular ejection fraction (LVEF) less than (<) 50 percent (%) as assessed after completion of induction treatment by either 2-dimensional echocardiogram or multiple-gated acquisition
* Clinically significant cardiovascular disease, including unstable angina, history of or active congestive heart failure of ≥ NYHA Grade 2, history of or ongoing serious cardiac arrhythmia requiring treatment (except for controlled atrial fibrillation and/or paroxysmal supraventricular tachycardia).
* Current uncontrolled hypertension with or without medication
* Current dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy
* Insulin-dependent diabetes
* Current known infection with HIV, HBV, or HCV (active infection or carriers)
* Requirement for concurrent use of the antiviral agent sorivudine (antiviral) or chemically related analogues, such as brivudine
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, or ulcerative colitis
* Known hypersensitivity to murine proteins

Exclusion Criteria for Participants in Cohort 4 (MP):

* Inability to swallow medications
* History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on most recent chest imaging (CT scan or MRI)
* Malabsorption condition that would alter the absorption of orally administered medications
* Amylase or lipase ≥ 1.5 times the upper limit of normal within 14 days prior to maintenance treatment initiation
* Serum albumin less than (<) 2.5 grams per deciliter (g/dL)
* LVEF < institutional lower limit of normal or < 50%, whichever is lower
* Poorly controlled hypertension
* Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage more than once every 28 days. Indwelling drainage catheters are allowed
* Unstable angina, new onset angina within last 3 months, myocardial infarction within last 6 months and current congestive heart failure ≥ NYHA Grade 2
* History of stroke, reversible ischemic neurological defect, or transient ischemic attack within 6 months prior to initiation of maintenance treatment
* History or evidence of intracranial hemorrhage or spinal cord hemorrhage
* Evidence of clinically significant vasogenic edema
* Any hemorrhage or bleeding event ≥ National Cancer Institute Common Terminology Criteria for Adverse Events Grade 3 within 28 days prior to initiation of maintenance treatment
* History or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for central serous retinopathy, retinal vein occlusion, or neovascular macular degeneration
* Positive HIV test
* Active HBV or HCV
* Active tuberculosis
* Severe infection within 4 weeks prior to start of maintenance treatment including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia; has signs or symptoms of significant infection or has received oral or IV antibiotics within 2 weeks prior to start of maintenance treatment.
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Administration of a live, attenuated vaccine within 4 weeks prior to start of study maintenance treatment or anticipation that such a live attenuated vaccine will be required during the study
* Prior treatment with CD137 agonists, anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Prior treatment with a mitogen-activated protein kinase/extracellular signal-regulated kinase (ERK) or ERK inhibitor
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or five half-lives of the drug, whichever is longer, prior to start of study maintenance treatment
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to start of study maintenance treatment, or requirement for systemic immunosuppressive medications during the trial.
* If receiving a RANKL inhibitor (for example, denosumab), unwilling to adopt alternative treatment such as (but not limited to) bisphosphonates, while receiving atezolizumab.
* Consumption of foods, supplements or drugs that are potent cytochrome P450 3A4 (CYP3A4) enzyme inducers or inhibitors ≤ 7 days before initiation of study maintenance treatment or expected concomitant use during maintenance treatment. These include St. John's wort or hyperforin (potent CYP3A4 enzyme inducer) and grapefruit juice (potent CYP3A4 enzyme inhibitor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2015-04-17 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (154):
- Argentina (3):
  - Hospital de Gastroenterologia Dr. Bonorino Udaondo ; Servicio de Oncología, Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Clínica Viedma, Viedma Rio Negro
- Belgium (5):
  - Institut Jules Bordet X, Brussels
  - Hospital Erasme, Brussels
  - UZ Leuven Gasthuisberg, Leuven
  - CHC MontLégia, Liège
  - AZ Delta (Campus Rumbeke), Roeselare
- University Clinical Center of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Brazil (7):
  - Hospital da Cidade de Passo Fundo; Centro de Pesquisa em Oncologia, Passo Fundo, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Faculdade de Medicina de Sao Jose do Rio Preto - FAMERP*X*, São José do Rio Preto, São Paulo
  - Instituto de Ensino e Pesquisa Sao Lucas - IEP, São Paulo, São Paulo
- Denmark (5):
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
  - Regionshospitalet Gødstrup; Kræftafdelingen, Herning
  - Rigshospitalet; Onkologisk Klinik, København Ø
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
  - Sygehus Syd Roskilde; Onkologisk/haematologisk ambulatorium, Roskilde
- Egypt (2):
  - National Cancer Institute, Cairo
  - Ain Shams University Hospital; Oncology, Cairo
- France (14):
  - Clinique Sainte Catherine, Avignon
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Hopital Augustin Morvan; Federation De Cancerologie, Brest
  - Chu Estaing; Chir Generale Digestive A Et B, Clermont-Ferrand
  - Hôpital Franco-Britannique- Fondation Cognacq-Jay; Cancerologie, Levallois-Perret
  - Hopital Claude Huriez; Medecine Interne Oncologie, Lille
  - Ch De Montbeliard;Chir Generale Digestive, Montbéliard
  - Hopital Caremeau; Gastro Enterologie, Nîmes
  - Hopital Saint Antoine; Oncologie Medicale, Paris
  - Hopital Haut Leveque, Pessac
  - Chu La Miletrie; Gastro Enterologie Endoscopies, Poitiers
  - ICANS, Strasbourg
  - Hopital Rangueil; Gastro Enterologie Et Nutrition, Toulouse
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif
- Germany (27):
  - Hämatologie Onkologie im Zentrum MVZ GmbH, Augsburg
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - DRK Kliniken Berlin Köpenick Darmzentrum, Berlin
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf; Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Krankenhaus Nordwest; Klinik f. Onkologie und Hämatologie, Frankfurt
  - PIOH PD Dr. R. Schnell ? Dr. H. Schulz ? Dr. M. Hellmann, Frechen
  - Klinik Fulda, Medizinisches Versorgungszentrum Osthessen GmbH, Fulda
  - Universitätsklinikum Hamburg-Eppendorf, Onkologisches Zentrum, Studienzentrale der II. Med. Klinik, Hamburg
  - Medizinische Hochschule Hannover; Zentrum Innere Medizin; Abt. Hämatologie u. Onkologie, Hanover
  - SLK-Kliniken Heilbronn GmbH; Klinik für Innere Medizin III; Schwerpunkt Häma./Onko./Palliativm., Heilbronn
  - Klinik der Ruhr-Uni Bochum; Marien-Hospital Herne, Herne
  - Gemeinschaftspraxis für Hämatologie und Onkologie, PD Dr. Bauer, Dr. Thiel, Lebach
  - Onkologische Gemeinschaftspraxis, Magdeburg
  - Klinikum Magdeburg gGmbH Klinik für Allgemein- und Viszeralchirurgie, Magdeburg
  - Universitätsklinikum Magdeburg Klinik für Gastroenterologie und Hepatologie, Mageburg
  - Kliniken Maria Hilf GmbH, Krankenhaus St. Franziskus, Mönchengladbach
  - Städt. Klinikum München GmbH Klinikum Neuperlach Klinik f.Hämatologie u.Onkologie, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Brüderkrankenhaus St. Josef, Paderborn
  - Studienzentrum Onkologie Ravensburg GbR; Onkologie Ravensburg, Ravensburg
  - Prosper-Hospital, Medizinische Klinik I, Recklinghausen
  - Krankenhaus Barmherziger Brüder; Klinik für Internistische Onkologie / Hämatologie, Regensburg
  - Klinikum am Steinenberg / Ermstalklinik, Reutlingen
  - Praxis für Hämatologie & Onkologie, Saarbrücken
  - MVZ für Hämatologie, Onkologie, Strahlentherapie und Palliativmedizin -; Klinik Dr. Hancken, Stade
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH; Haematologie/Onkologie, Trier
  - Klinikum Wetzlar-Braunfels, Klinik für Hämatologie/Onkologie und Palliativmedizin, Wetzlar
- Greece (7):
  - Agioi Anargyroi; 3Rd Dept. of Medical Oncology, Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - Uni Hospital of Ioannina; Oncology Dept., Ioannina
  - University Hospital of Patras Medical Oncology, Pátrai
  - Thermi Clinic; Oncology Clinic, Thermi Thessalonikis
  - Bioclinic Thessaloniki, Thessaloniki
  - Euromedical General Clinic of Thessaloniki; Oncology Department, Thessaloniki
- Italy (13):
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Oncologia, San Giovanni Rotondo, Apulia
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale; Oncologia Medica A, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - A.O. Universitaria Di Parma; Oncologia Medica, Parma, Emilia-Romagna
  - Istituto Regina Elena; Oncologia Medica A, Rome, Lazio
  - Policlinico Universitario "Agostino Gemelli"; U.O.C. Oncologia Medica, Rome, Lazio
  - Humanitas Gavazzeni;U.O. Oncologia Medica, Bergamo, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 1, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria Careggi;S.C. Oncologia Medica 1, Florence, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Prima, Padua, Veneto
  - A.O.U.I. VERONA-OSPEDALE POLICLINICO G.B. ROSSI BORGO ROMA;ONCOLOGIA MEDICA-d.U., Verona, Veneto
- Mexico (4):
  - Fundacion Rodolfo Padilla Padilla A.C., León, Guanajuato
  - Oaxaca Site Management Organization, Oaxaca City, Oaxaca
  - Cancerologia de Queretaro; Oncologia, Queretaro, Queretaro, Querétaro
  - Instituto Nacional de Cancerologia; Oncology, Mexico City
- Netherlands (7):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Ijsselland Ziekenhuis; Inwendige Geneeskunde, Capelle aan den IJssel
  - Deventer Ziekenhuis; Interne Geneeskunde, Deventer
  - Albert Schweitzer Ziekenhuis - loc Dordrecht, Dordrecht
  - Catharina ZKHS; Inwendige Geneeskunde Afd., Eindhoven
  - St. Antonius locatie Leidsche Rijn, Utrecht
  - Isala Klinieken, Zwolle
- Poland (2):
  - Szpital Uniwersytecki w Krakowie, Oddzia? Kliniczny Kliniki Onkologii, Krakow
  - Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie; Klinika Onkologii i Radioterapii,, Warsaw
- Portugal (2):
  - HUC; Servico de Oncologia Medica, Coimbra
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
- Russia (2):
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa, Bashkortostan Republic
  - Russian Oncology Research Center n.a. N.N. Blokhin Dpt of Clinical Pharmacology and Chemotherapy, Moscow, Moscow Oblast
- Institute for Oncology and Radiology of Serbia; Clinic for Medical Oncology, Belgrade, Serbia
- Slovakia (2):
  - Narodny Onkologicky Ustav; Oddelenie klinickej onkologie E, Bratislava
  - POKO Poprad; Department of Oncology, Poprad
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (26):
  - Hospital General Universitario de Elche; Servicio de Oncologia, Elche, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital de Donostia; Servicio de Oncologia Medica, Donostia / San Sebastian, Guipuzcoa
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Majadahonda, Madrid
  - Hospital de Navarra; Servicio de Oncologia, Navarra, Navarre
  - Hospital Univ. Central de Asturias; Servicio de Oncologia, Oviedo, Principality of Asturias
  - Complejo Hospitalario Nuestra Señora de la Candelaria; Servicio de Oncologia, Santa Cruz de Tenerife, Tenerife
  - Hospital General Univ. de Alicante; Servicio de Oncologia, Alicante
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Oncologia, Lleida
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga
  - Complejo Hospitalario de Orense; Servicio de Oncologia, Ourense
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa; Servicio de Oncologia, Zaragoza
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (2):
  - Skånes University Hospital, Skånes Department of Onclology, Lund
  - Karolinska Hospital; Oncology - Radiumhemmet, Stockholm
- Turkey (Türkiye) (6):
  - Acibadem University School of Medicine, Adana Hospital; General Surgery, Adana
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Istanbul Uni Capa Medical Faculty; Inst. of Oncology, Istanbul
  - Marmara Uni Faculty of Medicine; Medical Oncology, Istanbul
  - Ege Uni Medical Faculty Hospital; Oncology Dept, Izmir
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sihhiye/Ankara
- United Kingdom (11):
  - Aberdeen Royal Infirmary; Medical Oncology Dept, Aberdeen
  - Birmingham Heartlands Hospital, Birmingham
  - Broomfield Hospital; Oncology, Chelsmford
  - Castle Hill Hospital; The Queens Centre for Oncology and Haematology, Cottingham
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Royal Marsden Hospital; Dept of Med-Onc, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - Mount Vernon Hospital, Middlesex
  - Queen's Hospital, Romford
  - Southampton General Hospital; Medical Oncology, Southampton
  - Royal Marsden Hospital; Dept. of Medicine, Sutton

REFERENCES:
- [Derived] Ducreux M, Tabernero J, Grothey A, Arnold D, O'Dwyer PJ, Gilberg F, Abbas A, Thakur MD, Prizant H, Irahara N, Tahiri A, Schmoll HJ, Van Cutsem E, de Gramont A. Clinical and exploratory biomarker findings from the MODUL trial (Cohorts 1, 3 and 4) of biomarker-driven maintenance therapy for metastatic colorectal cancer. Eur J Cancer. 2023 May;184:137-150. doi: 10.1016/j.ejca.2023.01.023. Epub 2023 Feb 4. PMID 36921494

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants initially received study treatment during the Induction Phase. Next, participants within each cohort based on biomarker status were randomized to either an experimental arm or control arm per cohort in the Maintenance Phase. BRAFmut participants experiencing early disease progression during induction treatment had the option of proceeding immediately to receive second-line treatment and were followed during the study, but were not part of the Maintenance Phase study objectives.
Groups:
- Cohort 1: Induction Phase (IP): Included participants with v-raf murine sarcoma viral oncogene homolog B1 mutation positive (BRAFmut)/human epidermal growth factor receptor 2 negative (HER2-)/microsatellite stable (MSS)/rat sarcoma wild type (RASwt). All study participants received either eight 2-week cycles of 5-fluorouracil (5-FU)/ leucovorin calcium (LV) and oxaliplatin (FOLFOX) in combination with bevacizumab, or six 2-week cycles of FOLFOX in combination with bevacizumab, followed by two 2-week cycles of 5-FU/LV with bevacizumab during Induction Treatment.
- Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib: Participants with v-raf murine sarcoma viral oncogene homolog B1 mutation positive (BRAFmut)/human epidermal growth factor receptor 2 negative (HER2-)/microsatellite stable (MSS)/rat sarcoma wild type (RASwt) received 1600-2400 milligrams per square meter (mg/m^2) 5-FU via 46-hour intravenous (IV) infusion in combination with 400 mg/m^2 LV via 2-hour infusion on Day 1 of every 2-week cycle with 500 mg/m^2 cetuximab via infusion on Day 1 of every 2-week cycle and 960 milligrams (mg) vemurafenib twice daily (BID) by mouth.
- Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab: Per Investigator discretion, participants received fluoropyrimidine (5-FU/LV or capecitabine) at a dose and schedule per the Investigator's discretion in accordance with locally approved prescribing information and 5 mg/kg bevacizumab via 1-30 minute IV on Day 1 of every 2-week cycle.
- Cohort 2 (IP): Included participants with BRAFwt. All study participants received either eight 2-week cycles of 5-fluorouracil (5-FU)/ leucovorin calcium (LV) and oxaliplatin (FOLFOX) in combination with bevacizumab, or six 2-week cycles of FOLFOX in combination with bevacizumab, followed by two 2-week cycles of 5-FU/LV with bevacizumab during Induction Treatment.
- Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab: Participants with BRAFwt received fluoropyrimidine (1600-2400 mg/m^2 5-FU via 46-hour IV infusion in combination with 400 mg/m^2 LV via 2-hour infusion on Day 1 of every 2-week cycle or 1000 mg/m^2 twice-daily capecitabine BID by mouth on Days 1-14 every 2 weeks followed by a 1-week break) with 5 milligrams per kilogram (mg/kg) bevacizumab via 15-30 minute IV infusion on Day 1 of every 2-week cycle and 800 mg atezolizumab via 60-minute IV infusion on Day 1 of every 2-week cycle.
- Cohort 3 (IP): Included participants with human epidermal growth factor receptor 2 positive (HER2+). All study participants received either eight 2-week cycles of 5-fluorouracil (5-FU)/ leucovorin calcium (LV) and oxaliplatin (FOLFOX) in combination with bevacizumab, or six 2-week cycles of FOLFOX in combination with bevacizumab, followed by two 2-week cycles of 5-FU/LV with bevacizumab during Induction Treatment.
- Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab: Participants with human epidermal growth factor receptor 2 positive (HER2+) received 1000 mg/m^2 twice-daily capecitabine BID by mouth on Days 1-14 every 2 weeks followed by a 1-week break with trastuzumab by IV infusion on Day 1 of every 3-week treatment cycle at an initial loading dose of 8 mg/kg followed by 6 mg/kg for subsequent doses, and pertuzumab by IV infusion on Day 1 of each 3-week treatment cycle at an initial fixed loading dose of 840 mg followed by 420 mg for subsequent doses.
- Cohort 4 (IP): Included participants with HER2-/high microsatellite instability (MSI-H); HER2-/MSS/v-raf murine sarcoma viral oncogene homolog B1 wild type (BRAFwt); HER2-/MSS/BRAFmut/rat sarcoma mutation positive (RASmut). All study participants received either eight 2-week cycles of 5-fluorouracil (5-FU)/ leucovorin calcium (LV) and oxaliplatin (FOLFOX) in combination with bevacizumab, or six 2-week cycles of FOLFOX in combination with bevacizumab, followed by two 2-week cycles of 5-FU/LV with bevacizumab during Induction Treatment.
- Cohort 4 (MP): Cobimetinib,Atezolizumab: Participants with HER2-/high microsatellite instability (MSI-H); HER2-/MSS/v-raf murine sarcoma viral oncogene homolog B1 wild type (BRAFwt); HER2-/MSS/BRAFmut/rat sarcoma mutation positive (RASmut) received 60 mg cobimetinib orally for 3 weeks followed by a 1-week treatment break and atezolizumab at a fixed dose of 840 mg via 60-minute IV infusion on Day 1 of every 2-week cycle.
- Early Progressing BRAFmut Cohort: BRAFmut participants experiencing early disease progression during induction treatment had the option of proceeding immediately to receive second-line treatment with 5-FU/LV, cetuximab and vemurafenib if their primary tumor was MSS, or with a fluoropyrimidine (5-FU/LV or capecitabine), bevacizumab, and atezolizumab if their primary tumor was MSI-H. This cohort was followed during the study, but was not part of the Maintenance Phase study objectives.
Period: Induction Treatment
Arm/Group | Cohort 1: Induction Phase (IP) | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (IP) | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (IP) | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (IP) | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Early Progressing BRAFmut Cohort
Started | 93 | 0 | 0 | 635 | 0 | 0 | 6 | 0 | 0 | 310 | 0 | 0 | 0
Treated During Induction Phase | 93 | 0 | 0 | 632 | 0 | 0 | 6 | 0 | 0 | 309 | 0 | 0 | 0
Completed | 63 | 0 | 0 | 460 | 0 | 0 | 5 | 0 | 0 | 135 | 0 | 0 | 0
Not Completed | 30 | 0 | 0 | 175 | 0 | 0 | 1 | 0 | 0 | 175 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0 | 0 | 18 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 25 | 0 | 0 | 111 | 0 | 0 | 1 | 0 | 0 | 82 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 12 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0
Not completed — Non-Compliance | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Missing | 4 | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 54 | 0 | 0 | 0
Period: Maintenance Treatment Phase
Arm/Group | Cohort 1: Induction Phase (IP) | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (IP) | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (IP) | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (IP) | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Early Progressing BRAFmut Cohort
Started | 0 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 40 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 20 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 0 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 297 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 148 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 0 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 3 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 2 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 0 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 65 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 34 (Participants from IP Cohorts were randomized to the MP Cohorts based on bio-marker assessments.) | 0
Treated During Maintenance Phase | 0 | 40 | 18 | 0 | 293 | 143 | 0 | 3 | 2 | 0 | 64 | 34 | 0
Completed | 0 | 6 | 2 | 0 | 66 | 21 | 0 | 0 | 1 | 0 | 12 | 6 | 0
Not Completed | 0 | 34 | 18 | 0 | 231 | 127 | 0 | 3 | 1 | 0 | 53 | 28 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 15 | 12 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Not completed — Death | 0 | 29 | 16 | 0 | 188 | 107 | 0 | 1 | 1 | 0 | 46 | 19 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 15 | 4 | 0 | 1 | 0 | 0 | 3 | 3 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 7 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Not Treated | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Ended by Sponsor | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Early Disease Progression
Arm/Group | Cohort 1: Induction Phase (IP) | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (IP) | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (IP) | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (IP) | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Early Progressing BRAFmut Cohort
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Induction Phase (IP) | Cohort 2 (IP) | Cohort 3 (IP) | Cohort 4 (IP) | Total
Number analyzed (Participants) | 93 | 635 | 6 | 310 | 1044
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (12.0) | 60.9 (12.6) | 48.0 (7.7) | 60.1 (10.3) | 60.5 (11.9)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0
  Adults (18-64 years) | 58 | 351 | 6 | 199 | 614
  From 65-84 years | 35 | 279 | 0 | 110 | 424
  85 years and over | 0 | 5 | 0 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 247 | 4 | 123 | 423
  Male | 44 | 388 | 2 | 187 | 621
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 52 | 1 | 49 | 107
  Not Hispanic or Latino | 75 | 494 | 4 | 247 | 820
  Unknown or Not Reported | 13 | 89 | 1 | 14 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 9 | 0 | 14 | 24
  Asian | 5 | 15 | 0 | 16 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 10 | 0 | 5 | 15
  White | 76 | 539 | 6 | 264 | 885
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 11 | 62 | 0 | 9 | 82

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first occurrence of disease progression according to RECIST v1.1, or death from any cause, whichever occurs first. Progressive disease (PD) for target lesion: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/=5 mm. PD for non-target lesion: Unequivocal progression of existing non-target lesions.
Time Frame: From randomization until disease progression or death from any cause, up to 5 years
Population: Participants that were in the Maintenance Phase of the study, which included the experimental and control arms of Cohorts 1-4.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab
Number analyzed (Participants) | 40 | 20 | 297 | 148 | 3 | 2 | 65 | 34
months | 9.99 [7.72 to 12.55] | 11.60 [3.58 to 15.67] | 7.13 [6.14 to 8.41] | 7.36 [5.82 to 8.94] | 4.44 [3.55 to 14.69] | 4.04 [4.04 to 5.39] | 3.75 [3.42 to 3.91] | 7.79 [3.98 to 9.46]
Statistical Analysis 1: Comparison: Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib vs Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.872, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.50 to 1.82]
Statistical Analysis 2: Comparison: Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab vs Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.666, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.77 to 1.18]
Statistical Analysis 3: Comparison: Cohort 4 (MP): Cobimetinib,Atezolizumab vs Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.128, Log Rank; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.90 to 2.29]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization into the MTP to time of death from any cause.
Time Frame: From randomization until death from any cause, up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab
Number analyzed (Participants) | 40 | 20 | 297 | 148 | 3 | 2 | 65 | 34
months | 24.02 [16.07 to 34.00] | 21.73 [7.92 to 37.19] | 22.54 [20.04 to 26.87] | 22.24 [18.50 to 25.13] | NA [NA to 16.07] — not evaluable | 14.59 [NA to NA] — not evaluable | 22.60 [14.23 to 27.40] | 25.17 [15.90 to 32.59]
Statistical Analysis 1: Comparison: Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib vs Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.276, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.39 to 1.32]
Statistical Analysis 2: Comparison: Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab vs Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.076, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.64 to 1.02]
Statistical Analysis 3: Comparison: Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab vs Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.157, Log Rank
Statistical Analysis 4: Comparison: Cohort 4 (MP): Cobimetinib,Atezolizumab vs Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.415, Log Rank; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.73 to 2.14]

3. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: From baseline until end of study (up to 5 years)
Population: Safety population: all participants who received an intervention during the study.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1 Control: 5-FU/LV or Capecitabin, Bevacizumab; Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab: Per Investigator discretion, participants received fluoropyrimidine (5-FU/LV or capecitabine) at a dose and schedule per the Investigator's discretion in accordance with locally approved prescribing information and 5 mg/kg bevacizumab via 1-30 minute IV on Day 1 of every 2-week cycle.
Arm/Group | Cohort 1: Induction Phase (IP) | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control: 5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (IP) | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (IP) | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (IP) | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Early Progressing BRAFmut Cohort
Number analyzed (Participants) | 93 | 40 | 18 | 631 | 293 | 143 | 6 | 3 | 2 | 309 | 64 | 34 | 11
percentage of participants | 98.9 | 100 | 94.4 | 96.0 | 95.6 | 88.1 | 100 | 100 | 100 | 97.4 | 98.4 | 88.2 | 90.9

4. Secondary Outcome: Overall Response
Description: Calculated as the number of participants with a best overall response of CR or PR according to RECIST 1.1. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. OR= CR + PR.
Time Frame: From randomization until disease progression, up to 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Control(MP): 5-FU/LV or Capecitabin, Bevacizumab; Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab: Per Investigator discretion, participants received fluoropyrimidine (5-FU/LV or capecitabine) at a dose and schedule per the Investigator's discretion in accordance with locally approved prescribing information and 5 mg/kg bevacizumab via 1-30 minute IV on Day 1 of every 2-week cycle.
Arm/Group | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control(MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab
Number analyzed (Participants) | 40 | 20 | 297 | 148 | 3 | 2 | 65 | 34
Participants | 20 | 5 | 49 | 22 | 1 | 0 | 7 | 8
Statistical Analysis 1: Comparison: Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib vs Cohort 1 Control(MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.064, Chi-squared
Statistical Analysis 2: Comparison: Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab vs Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.658, Chi-squared
Statistical Analysis 3: Comparison: Cohort 4 (MP): Cobimetinib,Atezolizumab vs Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.093, Chi-squared

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with CR, PR, or stable disease (SD) at 16 weeks. Per RECIST v1.1, CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum on study. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline, or the appearance of one or more new lesions.
Time Frame: From randomization until disease progression, up to 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control(MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab
Number analyzed (Participants) | 40 | 20 | 297 | 148 | 3 | 2 | 65 | 34
Participants | 36 | 15 | 227 | 111 | 1 | 0 | 44 | 26
Statistical Analysis 1: Comparison: Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib vs Cohort 1 Control(MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.125, Chi-squared
Statistical Analysis 2: Comparison: Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab vs Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.739, Chi-squared
Statistical Analysis 3: Comparison: Cohort 4 (MP): Cobimetinib,Atezolizumab vs Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.362, Chi-squared

6. Secondary Outcome: Time to Treatment Response
Description: Calculated as the time from randomization to the first Occurrence of a documented Objective Response (CR or PR) determined according to RECIST 1.1. CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From randomization until disease progression or death from any cause, up to 5 years
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Groups:
- Cohort 1 Control(MP):5-FU/LV or Capecitabin, Bevacizumab; Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab: Per Investigator discretion, participants received fluoropyrimidine (5-FU/LV or capecitabine) at a dose and schedule per the Investigator's discretion in accordance with locally approved prescribing information and 5 mg/kg bevacizumab via 1-30 minute IV on Day 1 of every 2-week cycle.
Arm/Group | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control(MP):5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab
Number analyzed (Participants) | 40 | 20 | 297 | 148 | 3 | 2 | 65 | 34
months | 3.943 [1.18 to 29.70] | 5.552 [1.38 to 8.02] | 5.224 [1.22 to 26.74] | 4.616 [1.25 to 19.91] | 5.490 [5.490 to 5.490] | 0 [0 to 0] | 3.745 [1.77 to 14.92] | 2.530 [1.64 to 11.83]

7. Secondary Outcome: Duration of Response
Description: Defined as the time from the first assessment of CR or PR until disease progression or death from any cause, whichever occurs first. CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From first objective response until disease progression or death from any cause, up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control(MP):5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab
Number analyzed (Participants) | 40 | 20 | 297 | 148 | 3 | 2 | 65 | 34
months | 11.50 [7.66 to 21.49] | 8.74 [5.36 to 19.02] | 9.30 [5.55 to 11.30] | 7.59 [6.93 to 13.90] | 9.205 [9.205 to 9.205] | 0 [0 to 0] | 7.11 [1.48 to NA] — Upper value of the 95% CI cannot be calculated because it is above the maximum value observed. | 6.06 [2.20 to 7.33]
Statistical Analysis 1: Comparison: Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib vs Cohort 1 Control(MP):5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.421, Log Rank
Statistical Analysis 2: Comparison: Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab vs Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.495, Log Rank
Statistical Analysis 3: Comparison: Cohort 4 (MP): Cobimetinib,Atezolizumab vs Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab; Test type: Superiority; p = 0.357, Log Rank

8. Secondary Outcome: Percentage of Participants With Improvement and/or Stayed the Same on the Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score
Time Frame: From baseline until end of study (up to 5 years)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control(MP):5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab
Number analyzed (Participants) | 40 | 20 | 297 | 148 | 3 | 2 | 65 | 34
percentage of participants
  Improved | 10.0 | 5.0 | 10.4 | 5.4 | 0 | 0 | 7.7 | 5.9
  Improved or stayed the same | 75.0 | 85.0 | 76.7 | 82.5 | 100 | 100 | 63.1 | 79.4

ADVERSE EVENTS:
Time Frame: From baseline until end of study (up to 5 years)
Description: All-cause mortality was based on the intent-to-treat (ITT) population, which included all participants randomized in the study. Serious Adverse Events and Other Adverse Events were based on the safety population, which included all participants who received an intervention during the study.
Arm/Group | Cohort 1: Induction Phase (IP) | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib | Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 2 (IP) | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 3 (IP) | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Cohort 4 (IP) | Cohort 4 (MP): Cobimetinib,Atezolizumab | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab | Early Progressing BRAFmut Cohort
All-Cause Mortality (participants affected / at risk) | 25/93 | 29/40 | 16/20 | 111/635 | 188/297 | 107/148 | 1/6 | 1/3 | 1/2 | 82/310 | 46/65 | 19/34 | 10/11
Serious Adverse Events (participants affected / at risk) | 44/93 | 15/40 | 5/18 | 232/632 | 76/293 | 20/143 | 1/6 | 0/3 | 0/2 | 93/309 | 26/64 | 3/34 | 3/11
Other Adverse Events (participants affected / at risk) | 91/93 | 40/40 | 17/18 | 608/632 | 270/293 | 120/143 | 6/6 | 3/3 | 2/2 | 298/309 | 61/64 | 29/34 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Induction Phase (IP) (N=93) | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib (N=40) | Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab (N=18) | Cohort 2 (IP) (N=632) | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab (N=293) | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab (N=143) | Cohort 3 (IP) (N=6) | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab (N=3) | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab (N=2) | Cohort 4 (IP) (N=309) | Cohort 4 (MP): Cobimetinib,Atezolizumab (N=64) | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab (N=34) | Early Progressing BRAFmut Cohort (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 12 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 13 (14) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (3) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 10 (10) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 10 (10) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site thrombosis (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 14 (15) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 2 (2) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (2) | 0 (0) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 8 (11) | 2 (2) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Implant site dehiscence (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteral stent removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Choroidal effusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euthanasia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fournier's gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site impaired healing (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible cerebral vasoconstriction syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Induction Phase (IP) (N=93) | Cohort 1 (Maintenance Phase[MP]):5-FU/LV,Cetuximab,Vemurafenib (N=40) | Cohort 1 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab (N=18) | Cohort 2 (IP) (N=632) | Cohort 2 (MP):5-FU/LV or Capecitabine,Bevacizumab,Atezolizumab (N=293) | Cohort 2 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab (N=143) | Cohort 3 (IP) (N=6) | Cohort 3 (MP): Capecitabine,Trastuzumab,Pertuzumab (N=3) | Cohort 3 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab (N=2) | Cohort 4 (IP) (N=309) | Cohort 4 (MP): Cobimetinib,Atezolizumab (N=64) | Cohort 4 Control (MP): 5-FU/LV or Capecitabin, Bevacizumab (N=34) | Early Progressing BRAFmut Cohort (N=11)
Anaemia (Blood and lymphatic system disorders) | 20 (28) | 7 (10) | 1 (2) | 87 (114) | 21 (27) | 8 (13) | 1 (1) | 0 (0) | 0 (0) | 49 (62) | 8 (10) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 5 (6) | 1 (1) | 0 (0) | 40 (57) | 4 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 11 (14) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 22 (31) | 2 (2) | 1 (1) | 133 (220) | 12 (12) | 8 (17) | 0 (0) | 0 (0) | 0 (0) | 78 (123) | 7 (9) | 3 (4) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 0 (0) | 45 (67) | 10 (12) | 4 (10) | 0 (0) | 0 (0) | 0 (0) | 22 (45) | 4 (4) | 1 (5) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 18 (19) | 16 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 26 (34) | 24 (32) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 4 (5) | 4 (5) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 14 (17) | 4 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (7) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 28 (34) | 8 (10) | 1 (1) | 113 (152) | 39 (44) | 12 (15) | 1 (1) | 0 (0) | 0 (0) | 45 (56) | 12 (15) | 5 (5) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 12 (14) | 2 (2) | 3 (3) | 56 (69) | 18 (22) | 11 (15) | 0 (0) | 0 (0) | 0 (0) | 20 (21) | 5 (6) | 1 (1) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 23 (27) | 5 (6) | 0 (0) | 158 (235) | 38 (48) | 17 (26) | 2 (2) | 0 (0) | 1 (1) | 58 (74) | 7 (9) | 2 (2) | 1 (1)
Dental cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 52 (104) | 16 (43) | 4 (5) | 282 (539) | 78 (120) | 21 (36) | 4 (9) | 2 (5) | 0 (0) | 134 (276) | 40 (87) | 8 (11) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 7 (9) | 1 (1) | 1 (1) | 35 (43) | 10 (12) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 19 (19) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (8) | 2 (4) | 0 (0) | 17 (24) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 1 (1) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 2 (3) | 2 (3) | 0 (0) | 9 (9) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 7 (7) | 1 (1) | 1 (1) | 22 (24) | 5 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 53 (106) | 16 (23) | 0 (0) | 298 (589) | 64 (134) | 27 (41) | 2 (2) | 0 (0) | 0 (0) | 129 (246) | 17 (22) | 6 (22) | 3 (4)
Palatal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 18 (22) | 6 (6) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 24 (36) | 5 (6) | 3 (3) | 144 (225) | 35 (50) | 11 (19) | 0 (0) | 0 (0) | 0 (0) | 40 (52) | 1 (1) | 3 (3) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 23 (26) | 8 (8) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 29 (46) | 8 (12) | 1 (1) | 152 (243) | 39 (61) | 8 (11) | 1 (2) | 0 (0) | 0 (0) | 66 (101) | 13 (19) | 3 (9) | 4 (5)
Asthenia (General disorders) | 20 (32) | 5 (9) | 1 (2) | 115 (214) | 40 (58) | 12 (20) | 1 (1) | 0 (0) | 0 (0) | 63 (111) | 13 (18) | 3 (3) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 31 (50) | 9 (11) | 2 (2) | 247 (403) | 52 (77) | 23 (27) | 4 (6) | 1 (1) | 0 (0) | 87 (138) | 12 (20) | 7 (8) | 3 (3)
Influenza like illness (General disorders) | 5 (5) | 2 (2) | 0 (0) | 21 (22) | 9 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 1 (1) | 1 (1) | 1 (1)
Malaise (General disorders) | 2 (2) | 1 (1) | 0 (0) | 8 (9) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 16 (22) | 7 (8) | 2 (4) | 69 (90) | 20 (26) | 7 (9) | 3 (3) | 1 (1) | 0 (0) | 57 (72) | 4 (5) | 1 (1) | 2 (3)
Oedema peripheral (General disorders) | 9 (13) | 3 (6) | 0 (0) | 25 (25) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 16 (18) | 6 (8) | 1 (1) | 2 (3)
Pain (General disorders) | 3 (3) | 3 (3) | 0 (0) | 16 (16) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 19 (20) | 8 (8) | 1 (1) | 93 (144) | 32 (52) | 13 (14) | 2 (2) | 0 (0) | 0 (0) | 56 (76) | 20 (27) | 3 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (3) | 3 (3) | 0 (0) | 15 (15) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 0 (0) | 1 (2) | 17 (17) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 5 (6) | 3 (3) | 1 (1) | 16 (18) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 8 (10) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 8 (11) | 6 (8) | 0 (0) | 4 (5) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 42 (56) | 15 (21) | 10 (12) | 1 (1) | 1 (1) | 0 (0) | 15 (17) | 3 (4) | 1 (1) | 1 (1)
Onychomycosis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 6 (8) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 8 (22) | 5 (13) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (8)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 23 (23) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 3 (3) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 3 (4) | 2 (2) | 27 (40) | 12 (22) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 12 (13) | 2 (2) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 1 (1) | 1 (1) | 42 (52) | 12 (13) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 18 (25) | 7 (10) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (6) | 2 (3) | 0 (0) | 17 (28) | 10 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (17) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (7) | 2 (2) | 0 (0) | 34 (52) | 8 (14) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 17 (20) | 12 (13) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 4 (4) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 6 (9) | 1 (1) | 1 (1) | 35 (45) | 10 (13) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 20 (22) | 15 (15) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (3) | 1 (1) | 0 (0) | 19 (20) | 5 (5) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 12 (16) | 6 (6) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 4 (6) | 2 (3) | 1 (1) | 18 (24) | 8 (10) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 32 (40) | 31 (39) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 5 (8) | 4 (6) | 0 (0) | 13 (19) | 4 (4) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 5 (6) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 4 (4) | 3 (3) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (12) | 5 (7) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 4 (7) | 1 (1) | 0 (0) | 40 (74) | 6 (19) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 27 (37) | 6 (7) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 11 (12) | 4 (4) | 2 (2) | 64 (69) | 11 (12) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 30 (31) | 6 (6) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 10 (11) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (14) | 3 (7) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 16 (23) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (8) | 2 (4) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 20 (26) | 8 (10) | 0 (0) | 130 (171) | 24 (26) | 14 (15) | 2 (2) | 0 (0) | 0 (0) | 47 (55) | 11 (12) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 11 (11) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 1 (2)
Food craving (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 17 (23) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (3) | 1 (1) | 18 (37) | 5 (10) | 6 (10) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (20) | 3 (6) | 1 (1) | 68 (91) | 6 (7) | 8 (9) | 1 (1) | 1 (1) | 0 (0) | 16 (18) | 4 (4) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (9) | 6 (6) | 0 (0) | 9 (9) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 10 (10) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (48) | 18 (30) | 3 (5) | 74 (100) | 50 (67) | 8 (10) | 1 (1) | 0 (0) | 0 (0) | 19 (22) | 8 (8) | 3 (5) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (17) | 5 (5) | 2 (2) | 45 (59) | 22 (32) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 16 (17) | 5 (5) | 3 (3) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 10 (10) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 15 (15) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 10 (13) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (18) | 6 (8) | 1 (1) | 28 (34) | 15 (17) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 18 (23) | 5 (5) | 2 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (11) | 7 (10) | 0 (0) | 40 (50) | 13 (18) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 12 (14) | 5 (6) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 6 (11) | 4 (4) | 1 (2) | 29 (35) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 12 (12) | 4 (4) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 9 (11) | 4 (4) | 0 (0) | 59 (71) | 8 (8) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 21 (26) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (10) | 2 (2) | 0 (0) | 73 (179) | 24 (83) | 5 (15) | 1 (1) | 0 (0) | 0 (0) | 28 (50) | 6 (8) | 3 (5) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 10 (11) | 1 (1) | 0 (0) | 103 (145) | 18 (21) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | 57 (84) | 1 (2) | 5 (5) | 0 (0)
Neurotoxicity (Nervous system disorders) | 9 (15) | 3 (3) | 0 (0) | 22 (31) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 27 (46) | 3 (3) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 20 (29) | 4 (4) | 0 (0) | 93 (125) | 18 (21) | 10 (11) | 2 (2) | 0 (0) | 0 (0) | 43 (57) | 1 (1) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 3 (5) | 2 (3) | 0 (0) | 10 (11) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (12) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 26 (33) | 4 (5) | 1 (1) | 222 (357) | 32 (38) | 15 (16) | 3 (7) | 0 (0) | 0 (0) | 58 (91) | 3 (6) | 4 (4) | 0 (0)
Polyneuropathy (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 26 (35) | 6 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 9 (12) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 5 (7) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (7) | 1 (1) | 1 (1) | 19 (19) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 14 (14) | 2 (2) | 1 (1) | 38 (40) | 10 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 12 (13) | 3 (3) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1) | 20 (21) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (12) | 2 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 40 (56) | 17 (25) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 7 (12) | 1 (1) | 2 (4) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 5 (6) | 3 (3) | 77 (95) | 30 (39) | 9 (11) | 1 (1) | 0 (0) | 0 (0) | 27 (31) | 7 (7) | 3 (3) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1) | 1 (1) | 47 (61) | 15 (18) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 14 (14) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 2 (2) | 2 (2) | 47 (51) | 12 (12) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 20 (21) | 2 (2) | 1 (1) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (24) | 4 (4) | 1 (1) | 121 (157) | 23 (29) | 16 (20) | 3 (3) | 0 (0) | 2 (2) | 61 (70) | 6 (6) | 3 (4) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 20 (26) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 20 (27) | 6 (9) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (2) | 1 (1) | 19 (19) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (10) | 1 (1) | 2 (2) | 63 (64) | 8 (8) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 19 (19) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 12 (14) | 11 (13) | 0 (0) | 10 (11) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 20 (23) | 18 (20) | 2 (2) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (27) | 12 (16) | 3 (3) | 44 (54) | 18 (21) | 3 (6) | 1 (1) | 1 (1) | 0 (0) | 20 (20) | 6 (6) | 1 (1) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 11 (19) | 8 (11) | 1 (4) | 21 (22) | 11 (12) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (4)
Nail ridging (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 (19) | 5 (5) | 4 (5) | 98 (147) | 44 (66) | 25 (40) | 4 (7) | 3 (6) | 0 (0) | 19 (19) | 1 (1) | 3 (3) | 2 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 10 (11) | 9 (10) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (10) | 5 (5) | 2 (2) | 34 (42) | 20 (25) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 16 (26) | 7 (14) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 20 (24) | 13 (17) | 0 (0) | 43 (52) | 24 (30) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 38 (46) | 28 (33) | 0 (0) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (4) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 8 (12) | 7 (11) | 0 (0) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Skin toxicity (Skin and subcutaneous tissue disorders) | 6 (9) | 4 (7) | 0 (0) | 4 (5) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 8 (14) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (5) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 16 (21) | 1 (1) | 1 (1) | 170 (244) | 49 (70) | 15 (19) | 1 (1) | 0 (0) | 0 (0) | 62 (79) | 3 (4) | 5 (7) | 1 (1)
Hypotension (Vascular disorders) | 8 (8) | 4 (4) | 0 (0) | 10 (10) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 3 (3) | 0 (0) | 2 (2)
Auditory meatus external erosion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 9 (11) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 19 (21) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 3 (3) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 17 (22) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 25 (27) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 7 (8) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 13 (17) | 1 (1) | 0 (0) | 67 (108) | 7 (11) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 28 (42) | 2 (2) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 29 (43) | 5 (6) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 16 (20) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 7 (9) | 4 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Taste disorder (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 13 (13) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 12 (13) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 8 (12) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 3 (3) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Phlebitis (Vascular disorders) | 2 (3) | 1 (2) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 7 (8) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT02291289/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT02291289/SAP_001.pdf